CLINICAL TRIAL: NCT05446883
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate QL1706 Plus Paclitaxel-Cisplatin/Carboplatin With or Without Bevacizumab for the First-Line Treatment of Persistent, Recurrent or Metastatic Cervical Cancer
Brief Title: QL1706 Plus Chemotherapy±Bevacizumab for the First-Line Treatment of Persistent, Recurrent or Metastatic Cervical Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL1706-301
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: METASTATIC CERVICAL CANCER
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706+chemotherapy± bevacizumab (Experimental): QL1706 (5 mg/kg) + paclitaxel (175 mg/m2) + cisplatin (50 mg/m2)/carboplatin (AUC 5) ± bevacizumab (15 mg/kg)
  Interventions: Drug: QL1706; Drug: Paclitaxel injection; Drug: Cisplatin/Carboplatin
- Placebo+chemotherapy± bevacizumab (Placebo Comparator): Placebo + paclitaxel (175 mg/m2) + cisplatin (50 mg/m2)/carboplatin (AUC 5) ± bevacizumab (15 mg/kg)
  Interventions: Drug: Placebo; Drug: Paclitaxel injection; Drug: Cisplatin/Carboplatin

INTERVENTIONS:
Drug: QL1706 — Intravenous Infusion
  Arms: QL1706+chemotherapy± bevacizumab
Drug: Placebo — Intravenous Infusion
  Arms: Placebo+chemotherapy± bevacizumab
Drug: Paclitaxel injection — Intravenous Infusion
Drug: Cisplatin/Carboplatin — Intravenous Infusion

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multicenter phase III clinical study in 498 patients with persistent, recurrent or metastatic cervical cancer.Experimental: QL1706 + Chemotherapy (Paclitaxel-cisplatin/Carboplatin) ± Bevacizumab; Control group: placebo + chemotherapy (paclitaxel-cisplatin/carboplatin) ± bevacizumab

DETAILED DESCRIPTION:
Subjects must provide sufficient archival or newly obtained tumor tissue samples to determine PD-L1 expression level to be eligible for screening.During the screening phase, eligible subjects will be stratified by use of bevacizumab (yes vs no), prior concurrent chemoradiation therapy (yes vs no), and PD- L1 level (CPS < 1 vs 1 ≤ CPS < 10 vs CPS ≥ 10) and randomized 1:1 into the experimental or control arm.Experimental: QL1706 + Chemotherapy (Paclitaxel-cisplatin/Carboplatin) ± Bevacizumab;Control group: placebo + chemotherapy (paclitaxel-cisplatin/carboplatin) ± bevacizumab

ELIGIBILITY:
Inclusion Criteria:

* The subject fully understood and voluntarily signed the informed consent form.
* Histologically confirmed cervical cancer.
* At least one measurable tumor lesion by CT or MRI according to RECIST 1.1 criteria.
* All subjects must provide archived or freshly obtained tumor tissue samples, approximately 7 (minimum of 5) unstained FFPE pathology slides (preferably newly obtained tumor tissue samples) within 5 years prior to randomization.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected survival ≥ 12 weeks.
* Adequate level of vital organ function

Exclusion Criteria:

* Previously received immunotherapy, including immune checkpoint inhibitory antibodies (such as: anti-PD-1, PD-L1, CTLA-4 antibodies, etc.), immune checkpoint agonistic antibodies (such as: anti-ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), and immune cell therapy; previously received VEGF/VEGFR inhibitors, such as bevacizumab, ramucirumab, abercept and tyrosine kinase inhibitors.
* Systemic infection or other serious infection requiring intravenous antibiotics for 7 days before randomization, or unexplained fever > 38.5℃ during screening or before enrollment (except fever caused by tumor, as judged by the investigator)
* Within two weeks before randomization, there is a need for systemic use of corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive drugs (such as cyclophosphamide, azathioprine, methotrexate, thalidomide, TNF-α inhibitors, etc.) treatment of the disease; Topical corticosteroids, nasal sprays, and inhaled steroids are allowed. Systemic corticosteroids are permitted for the prevention of contrast allergy。
* Systemic treatment with immunomodulatory drugs (such as thymosin, lentinan, interferon, interleukin, etc.) within two weeks before randomization

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS by BICR based on RECIST v1.1 | Informed consent until disease progression or death, which ever occurs first (up to approximately 24 months)
  PFS by BICR based on RECIST v1.1
OS | From date of randomization until the date of death from any cause, whichever came first, assessed up to 2 years
  OS

SECONDARY OUTCOMES:
PFS and 12-month PFS rate assessed by investigator based on RECIST v1.1 criteria | Informed consent until disease progression or death, which ever occurs first (up to approximately 24 months
  PFS and 12-month PFS rate assessed by investigator based on RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Liaoning Cancer Hospital, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: No
Involves subject privacy and does not intend to share

REFERENCES:
- [Derived] Zhao Y, Ma Y, Zang A, Cheng Y, Zhang Y, Wang X, Chen Z, Qu S, He J, Chen C, Jin C, Zhu D, Li Q, Liu X, Su W, Ba Y, Hao Y, Chen J, Zhang G, Qu S, Li Y, Feng W, Yang M, Liu B, Ouyang W, Liang J, Yu Z, Kang X, Xue S, Yang G, Yan W, Yang Y, Liu Z, Peng Y, Fanslow B, Huang X, Zhang L, Zhao H. First-in-human phase I/Ib study of QL1706 (PSB205), a bifunctional PD1/CTLA4 dual blocker, in patients with advanced solid tumors. J Hematol Oncol. 2023 May 8;16(1):50. doi: 10.1186/s13045-023-01445-1. PMID 37158938